CLINICAL TRIAL: NCT02547909
Title: The Application of Probe-based Confocal Laser Endomicroscopy in the Diagnosis of Deep Endometriosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Ofir Harnoy MD (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Ofir Harnoy MD, Staff physician, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2146-15-SMC
Record Dates: First submitted 2015-08-31; First posted 2015-09-11 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Bowel Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study group (Experimental): a probe-based Confocal Laser Endomicroscopy examination will be done using a standard recto-sigmoidoscopy, in women suffering from endometriosis who are referred for a TRUS examination as part of a suspected deep endometriosis diagnostic workup. pCLE images will be compared to normal bowel mucosa.
  Interventions: Procedure: probe-based Confocal Laser Endomicroscopy; Device: Cellvizio; Drug: fluorescein 10%

INTERVENTIONS:
Procedure: probe-based Confocal Laser Endomicroscopy — Eligible women will be offered to undergo pCLE examination. Conscious sedation will be offered to all patients, who will choose to receive it or not. pCLE will be done using a standard gastroscope, reaching a distance of 25 cm from the anus, to the level of the rectosigmoid angle.
  At this point, 2.5 ml fluorescein 10% will be injected. The pCLE probe (GastroFlex-UHD probe, Mauna Kea tech, Paris, France) will be inserted through the endoscope working channel and images will be recorded from areas suspected of harboring an endometriotic tissue.
  Other Names: Cellvizio
Device: Cellvizio
Drug: fluorescein 10%

SUMMARY:
Endometriosis is defined as the presence of endometrial glands and stroma outside of the uterus.Endometriosis affects 5%-15% of women in the reproductive age. Deep endometriosis is mostly defined as a single endometrial nodule, located in the vesico-uterine fold or close to the distal 20 cm of the large bowel. Current guidelines recommends that laparoscopy with histology should be done to diagnose endometriosis. Probe-based confocal laser endomicroscopy (pCLE) has been used as a GI tract endoscopy additive tool in recent years, providing in-vivo cellular-level imaging, a concept known as "optical biopsy". considering the rectal bleeding that occurs in patients suffering from bowel endometriosis, usually with a normal mucosa seen at standard endoscopy (personal data), we hypothesized that there might be histological architectural changes in the vessels or the mucosa/sub mucosa in bowel endometriosis.

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial glands and stroma outside of the uterus, most commonly over the ovaries, fallopian tubes, bladder, recto-sigmoid colon and the uterine myometrium.Endometriosis affects 5%-15% of women in the reproductive age causing pelvic or abdominal pain, infertility and occasionally rectal bleeding (if involving the bowel). Deep endometriosis is mostly defined as a single endometrial nodule, usually larger than 1 cm which is located in the vesico-uterine fold or close to the distal 20 cm of the large bowel. Those lesions usually infiltrate at least 5 mm into the tissue involved. The gold standard of diagnosis is histological proven endometriosis, usually obtained during explorative laparoscopy. Other imaging tests that aid in the diagnosis are trans-vaginal or trans-rectal sonography (TRUS), MRI & CT. Current guidelines recommends that laparoscopy with histology should be done to diagnose endometriosis. Negative (normal) laparoscopy is highly accurate in excluding endometriosis, but a positive laparoscopy (i.e. with macroscopic findings) without biopsy has a limited value. In practice, many clinicians refrain from taking biopsies due-to the risk of bowel surgery, particularly on an un-prepared bowel. Probe-based confocal laser endomicroscopy (pCLE) has been used as a GI tract endoscopy additive tool in recent years, providing in-vivo cellular-level imaging, a concept known as "optical biopsy". considering the rectal bleeding that occurs in patients suffering from bowel endometriosis, usually with a normal mucosa seen at standard endoscopy (personal data), we hypothesized that there might be histological architectural changes in the vessels or the mucosa/sub mucosa in bowel endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis

Exclusion Criteria:

* Unable or unwilling to give and sign an informed consent
* Allergy to fluorescein
* Colitis
* Critical illness
* Pregnancy
* Malignancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
recognizing unique pCLE images for endometriosis | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Har-Noy, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel